CLINICAL TRIAL: NCT06408766
Title: Investigating the Short and Long-term Effects of Smartphone Use on the Masseter Muscle
Brief Title: Investigating the Effects of Smartphone Use on the Masseter Muscle
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, PhD, Bandırma Onyedi Eylül University
Other Study IDs: 2024-26
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-05

CONDITIONS: Smartphone Addiction; Masseter Muscle Hypertrophy; Masseter Muscle Spasm
Keywords: Smartphone Addiction; masseter; thenar
MeSH Terms: conditions — Internet Addiction Disorder; Masticatory Muscles, Hypertrophy of; Trismus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study was to determine the short- and long-term effects of smartphone use on the masseter muscle. In the short term, to investigate whether repetitive thumb movements during phone use will cause a spontaneous muscle activation and/or tenderness in the masseter muscle; in the long term, to investigate the relationship between strength change and tenderness of the tenar and masseter muscles depending on the intensity and duration of phone use.

DETAILED DESCRIPTION:
A total of 120 healthy university students aged 18-30 years at Bandırma Onyedi Eylül University will be included in our study. Descriptive data form, Smartphone Addiction Scale - Short Form, Edinburg Hand Preference Inventory, pressure pain threshold, muscle activity, lateral grip strength, hand grip strength will be evaluated in the participant students.

ELIGIBILITY:
Inclusion Criteria:

* Smartphone users students between the ages of 18-30 years
* Students whose voluntary informed consent was obtained

Exclusion Criteria:

* Individuals undergoing masseter botox application
* Individuals diagnosed with TMJ disorder and/or bruxism
* Individuals with musculoskeletal problems with evidence of a systemic, specific pathologic condition such as fracture of the hand, finger, upper extremity and/or TMJ, rheumatoid disease
* Individuals who have undergone any surgical operation related to hand, finger, upper extremity and/or TMJ problem
* Individuals with less than 6 months of physiotherapy and rehabilitation services related to hand, finger, upper extremity and/or TMJ
* Individuals with facial paralysis
* Individuals with diagnosed psychiatric illness.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Smartphone Addiction Scale-Short Form | 4 months
  In our study, the Smartphone Addiction Scale-Short Form will be filled out to evaluate the intensity of smartphone use of students, and the daily duration of smartphone use will be recorded. This scale consists of 10 6-point Likert-type items used to measure the risk of smartphone addiction. Scores on the scale range from 10-60, with an increase in score indicating an increased risk for smartphone addiction. The cut-off score of the scale was determined as 31 for men and 33 for women in the Korean sample.
Edinburg Hand Preference Inventory | 4 months
  Edinburg Hand Preference Inventory will be used to determine the dominant hand in our study. This scale asks which hand is used while performing 10 activities such as "writing", "drawing", "brushing teeth", "holding a fork (while eating)". For each activity; left hand preference is -10 points, right hand preference is +10 points and both hand preference is 0 points. After hand preference for all activities, the highest score that individuals can get is +100 and the lowest score is -100. A "negative" score is in favor of "left-handedness" and a "positive" score is in favor of "right-handedness". According to this scoring, individuals with a score between "+40 and +100" are recorded as "right-handed", individuals with a score between "-30 and +30" as "two-handed", and individuals with a score between "-100 and -40" as "left-handed".
Pressure Pain Threshold Assessment | 4 months
  In our study, pressure pain threshold measurement of the dominant and non-dominant side masseter and tenar muscles before and after the activity will be evaluated with Baseline manual algometer (2.5 kg-11 lb).
Muscle Activation Measurement | 4 months
  In our study, a four-channel Neurotrac Myoplus Pro 4 EMG Biofeedback device will be used for superficial electromyographic (EMG) measurements of the masseter muscle. The results of electromyographic activity will be presented as both mean data (microvolts) and normalized mean data (%MVC- Maximum Voluntary Contraction). The mean, minimum and peak contraction values of the activation will be recorded, the variability of the activation produced will be evaluated with the Inter Quantile Range (IQR). The average muscle activations that will occur in the muscle will be used as %MVC.
Hand Grip Strength Assessment | 4 months
  Hand grip strength will be measured with 'Saehan Hydraulic Hand Dynamometer'. A total of three measurements will be made for each hand with a 15 s break between each measurement of the extremity and the average of the three measurements will be taken. Test results will be recorded in kilograms.
Finger Lateral Grip Strength Assessment | 4 months
  Hand grip strength will be measured with 'Saehan Hydraulic pinch gauge'. Three measurements will be made for each hand in total with a 30-second break between each measurement and the average of the three measurements will be recorded in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylul University, Balıkesir, Bandirma, Turkey (Türkiye)